CLINICAL TRIAL: NCT06255236
Title: An Accuracy of Bispectral Index Monitoring in an Alternative Nasal Position Compared With Standard Frontal Position in Pediatric Patients Under General Anesthesia With Sevoflurane
Brief Title: Pediatric Frontal and Nasal Bispectral Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Si 785/2023
Record Dates: First submitted 2024-01-15; First posted 2024-02-13 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: BIS
Keywords: Pediatric anesthesia; Intraoperative care; Intraoperative neurophysiological monitoring
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- BIS (Experimental): The patients will receive both standard frontal and nasal BIS monitoring during general anesthesia.
  Interventions: Device: Bispectral index (BIS)

INTERVENTIONS:
Device: Bispectral index (BIS) — * All patient will receive standard monitoring (EKG, Blood pressure, pulse oximetry), and BIS transducer placement at standard frontal area before anesthesia.
  * Sedative medication can be given as appropriate.
  * Anesthesia induction by inhalation induction with sevoflurane (if intravenous line not presented) or intravenous induction with thiopental 5-6 mg/kg IV
  * Other medication including fentanyl 1 mcg/kg IV and cisatracurium 0.1-0.2 mg/kg IV will be given and the patient will be intubated.
  * The second BIS will be installed on the bridge of the nose and temporal on the same side as frontal BIS.
  * The patient will be maintained with sevoflurane and other anesthetic drugs as appropriate, adjusted per frontal BIS (40-60).
  * The frontal BIS and the nasal BIS will be measured until the endotracheal tube is being removed. If the patient has moved until it was impossible to measure the BIS or has any necessity to cancel the BIS measurement. The BIS measurement can be stopped.

SUMMARY:
To compare the accuracy of frontal versus nasal BIS monitoring in pediatric patients under general anesthesia.

DETAILED DESCRIPTION:
Standard position of frontal bispectral index (BIS) may not be available in some operations that frontal area is occupied by surgical field. This prospective cohort study aims to compare the accuracy of the BIS between an alternative position across the nasal area with the standard frontal BIS position in pediatric patients undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing general anesthesia
* American Society of Anesthesiologists physical status 1-3

Exclusion Criteria:

* Patients with neurological diseases
* Patients who are using anticonvulsant drugs
* Patients who is expected to be intubated and return to the pediatric intensive care unit
* Patients undergoing head and face surgery
* Patients undergoing surgery in the prone position
* Patients who have contraindications to sevoflurane, thiopental, fentanyl, and cisatracurium

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
bispectral index (BIS) value | 5 hours
  BIS is a processed electroencephalogram (range from 0-100), the optimal value of BIS during general anesthesia is 40-60. We aim to define the differences between standard frontal BIS and nasal BIS using Bland-Altman analysis.

SECONDARY OUTCOMES:
signal quality index (SQI) | 5 hours
  SQI (range from 0-100) determines the quality of signal of the primary outcome (BIS). We aim to define the differences of SQI of BIS between standard frontal and nasal positions.
electromyography (EMG) | 5 hours
  EMG (range from 0-100) reports the interference of muscle activity on quality of the primary outcome (BIS). We aim to define the differences of EMG between standard frontal and nasal positions.

CONTACTS AND LOCATIONS:
Overall Officials: Taniga Kiatchai, MD., Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson P, Nelson JA, Chen AJ, Kofke WA. An alternative position for the BIS-Vista montage in frontal approach neurosurgical cases. J Neurosurg Anesthesiol. 2013 Apr;25(2):135-42. doi: 10.1097/ANA.0b013e31826ca3a0. PMID 23456030